CLINICAL TRIAL: NCT00893490
Title: Ahmed Glaucoma Valve Alone,With Amniotic Membrane or With MMC for Treatment of Refractory Glaucoma
Brief Title: Ahmed Glaucoma Valve Alone, With Amniotic Membrane or With Mitomycin C (MMC) for Treatment of Refractory Glaucoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Ophthalmic Research Center
Purpose: Treatment
Other Study IDs: 8756
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2009-05-06 (Estimated); Status verified 2009-05

CONDITIONS: Refractory Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ahmed Glaucoma Valve (AGV) alone (Experimental)
  Interventions: Device: Ahmed Glaucoma Valve (AGV)
- AGV plus MMC (Experimental)
  Interventions: Device: Ahmed Glaucoma Valve (AGV); Drug: Mitomycin C (MMC)
- AGV plus amniotic membrane coverage (Experimental)
  Interventions: Device: Ahmed Glaucoma Valve (AGV); Procedure: amniotic membrane coverage

INTERVENTIONS:
Device: Ahmed Glaucoma Valve (AGV) — AGV implantation
Drug: Mitomycin C (MMC) — 3 minute MMC application
  Arms: AGV plus MMC
Procedure: amniotic membrane coverage — single layer coverage of amniotic membrane
  Arms: AGV plus amniotic membrane coverage

SUMMARY:
This randomized, controlled trial (RCT) compares the efficacy and safety of Ahmed Glaucoma Valve (AGV) implantation alone, with 3 minutes MMC application or with a single layer coverage of amniotic membrane. Outcomes include intraocular eye pressure (IOP), postoperative glaucoma medication and complications. AGV implantation site will be superior or inferior based on indication and these groups will be randomized separately.

ELIGIBILITY:
Inclusion Criteria:

* patients with refractory glaucoma

Exclusion Criteria:

* children under 7 years old
* adults above 75 years old
* uncooperative patients
* patients underwent the operation for second time
* patients with major operation with AGV

Ages: 7 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Tehran Province, Iran